CLINICAL TRIAL: NCT00579059
Title: A Randomized Data Collection of the Maxim® Knee System With Removable Molded Polyethylene Tibia and the Regular Maxim® Knee System
Brief Title: Maxim® Knee Pop-Top® Tibia vs. Regular Maxim® Knee Tibia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study sponsor canceled the study.
Sponsor: Biomet Orthopedics, LLC (Industry)
Responsible Party: Sponsor
Organization: Zimmer Biomet (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 62-U-007
Record Dates: First submitted 2007-12-17; First posted 2007-12-21 (Estimated); Results first posted 2009-07-07 (Estimated); Last update posted 2017-07-17 (Actual); Status verified 2017-06

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis; Traumatic Arthritis
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): Maxim® Pop-Top® Tibia
  Interventions: Device: Maxim® Knee System with Removable Molded Polyethylene Tibia
- 2 (Other): Maxim® Regular Tibia
  Interventions: Device: Regular Maxim® Knee System

INTERVENTIONS:
Device: Maxim® Knee System with Removable Molded Polyethylene Tibia — Used for total knee replacements
  Other Names: Maxim® Pop-Top® Tibia
  Arms: 1
Device: Regular Maxim® Knee System — Used for total knee replacements
  Other Names: Modular Tibia
  Arms: 2

SUMMARY:
The purpose of this prospective clinical data collection is to compare the outcomes of two different tibial bearings: the Maxim® Pop-Top® Tibia and Maxim® Modular Tibia.

DETAILED DESCRIPTION:
The purpose of this prospective clinical data collection is to document and compare the performance and clinical outcomes between the Maxim® Knee System with Removable Molded Poly Tibia and the Maxim® Knee System with Modular Tibial Bearing as two treatment groups.

FDA has cleared these devices via Premarket Notification 510(k)'s K991753, K984623, K993159, K010027. The data gathered will be collated and used to provide feedback to designing engineers, support marketing efforts and answer potential questions from reimbursement agencies.

ELIGIBILITY:
Inclusion Criteria:

Identical to the indications stated in the FDA approved labeling for the device (cleared in 510(k) K991753,

K984623, K993159, K010027). These indications are stated below:

* Painful and disabled knee joint resulting from osteoarthritis, rheumatoid arthritis, traumatic arthritis where one or more compartments are involved.
* Correction of varus, valgus, or posttraumatic deformity.
* Correction or revision of unsuccessful osteotomy, arthrodesis, or failure of previous joint replacement procedure.

Patient selection factors to be considered include:

* need to obtain pain relief and improve function,
* ability and willingness of the patient to follow instructions, including control of weight and activity level,
* a good nutritional state of the patient,
* the patient must have reached full skeletal maturity.
* Porous coated knee joint replacement prostheses have not been approved for non-cemented applications in the United States.

Exclusion Criteria:

Identical to the contraindications stated in the FDA approved labeling for the device (cleared in 510(k) K991753, K984623, K993159, K010027's). These contraindications are stated below:

Absolute contraindications include:

* infection,
* sepsis
* osteomyelitis.

Relative contraindications include:

* uncooperative patient or patient with neurologic disorders who are incapable of following directions,
* Osteoporosis,
* metabolic disorders which may impair bone formation,
* osteomalacia,
* distant foci of infections which may spread to the implant site,
* rapid joint destruction, marked bone loss or bone resorption apparent on roentgenogram,
* vascular insufficiency, muscular atrophy, neuromuscular disease,
* incomplete or deficient soft tissue surrounding the knee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2004-05; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Russell Wagner, MD, Principal Investigator — Harris Methodist Hospital
Locations (1):
- Biomet Orthopedics, LLC, Warsaw, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited by the investigator.
Pre-assignment Details: There were no pre-assignment details to report.
Groups:
- Maxim® Pop-Top® Tibia: tibia with removable polyethylene
- Maxim® Regular Tibia: Tibia with Modular Polyethylene
Period: Overall Study
Arm/Group | Maxim® Pop-Top® Tibia | Maxim® Regular Tibia
Started | 21 (Enrollment was incomplete due to study cancellation.) | 10 (Enrollment was incomplete due to study cancellation.)
Immediate Post-Op | 20 (1 Patient didn't return for follow-up.) | 9 (1 Patient didn't return for follow-up.)
6 Months | 11 (10 Patients didn't return for follow-up.) | 4 (6 patients didn't return for follow-up.)
1 Year | 8 (13 patients didn't return for follow-up.) | 3 (7 patients didn't return for follow-up.)
3 Years | 0 (Incomplete due to study closure at 1-year of follow-up.) | 0 (Incomplete due to study closure at 1-year of follow-up.)
5 Years | 0 (Incomplete due to study closure at 1-year of follow-up.) | 0 (Incomplete due to study closure at 1-year of follow-up.)
Completed | 0 (No Patients completed through 5 years due to study closure at 1-year of follow-up.) | 0 (No Patients completed through 5 years due to study closure at 1-year of follow-up.)
Not Completed | 21 | 10
Not completed — Study Canceled at 1 Year | 21 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Maxim® Pop-Top® Tibia | Maxim® Regular Tibia | Total
Number analyzed (Participants) | 21 | 10 | 31
Age, Continuous [Mean (Full Range); unit: years] | 68 (8) [53 to 82] | 62 (6) [54 to 75] | 65 [53 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 5 | 22
  Male | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  United States | 21 | 10 | 31.0

OUTCOME MEASURES:

1. Primary Outcome: Knee Society Function Score
Description: The function score is detailed below as a Range; 100 being the highest score, and 0 being the lowest score. 90-100 is considered "Excellent," 60-89 is considered "Good," 30-59 is considered "fair," and 0-29 is considered "poor."
Time Frame: 1 Year
Population: This population represents patients that returned for follow-up at 1-year post-op per protocol.
Measure: Number; unit: knees
Arm/Group | Maxim® Pop-Top® Tibia | Maxim® Regular Tibia
Number analyzed (Participants) | 8 | 3
knees
  90-100 | 6 | 2
  60-89 | 2 | 1
  30-59 | 0 | 0
  0-29 | 0 | 0

2. Secondary Outcome: Range of Motion - Flexion
Description: This represents how far the patients were able to flex the knee in the clinic at 1-year.
Time Frame: 1 Year
Population: This population represents patients that returned for follow-up at 1-year post-op per protocol.
Measure: Mean (Full Range); unit: degrees
Arm/Group | Maxim® Pop-Top® Tibia | Maxim® Regular Tibia
Number analyzed (Participants) | 8 | 3
degrees | 118 [100 to 130] | 113 [105 to 120]

ADVERSE EVENTS:
Time Frame: Not applicable - no adverse events were reported.
Arm/Group | Maxim® Pop-Top® Tibia | Maxim® Regular Tibia
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/10
Other Adverse Events (participants affected / at risk) | 0/21 | 0/10

LIMITATIONS AND CAVEATS:
Study was terminated after enrollment failed to produce sufficient data to be analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Biomet owns copyright to database.